CLINICAL TRIAL: NCT06239168
Title: The Effect of Citrus Extract on Sleep and Mental Wellbeing
Brief Title: Citrus Extract, Sleep and Mental Wellbeing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: BioActor (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-012
Record Dates: First submitted 2023-12-14; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — grapefruit seed extract; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citrus extract (Experimental): Daily Citrus extract supplementation for 8 weeks.
  Interventions: Dietary Supplement: Citrus extract
- Control (Placebo Comparator): Daily Maltodextrin supplementation for 8 weeks.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Citrus extract — As described in experimental arm
  Arms: Citrus extract
Dietary Supplement: Maltodextrin — As described in comparator arm
  Arms: Control

SUMMARY:
This is a randomized, double-blind, placebo-controlled, cross-over trial investigating the effects of daily administration of citrus extract on sleep and mental wellbeing.

DETAILED DESCRIPTION:
Based on epidemiological data, a substantial number of people report to have sleeping problems. This is of major concern, as poor sleep quality has been associated with impaired mental and physical health. Several pre-clinical studies have shown promising results, but evidence from human studies is still limited. Therefore, the aim of the present study is to investigate the effect of a citrus extract on sleep and mental wellbeing in healthy subjects with (minor) sleep disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with (minor) sleep disturbance
* Age 40-70 years
* BMI 18.5 - 30 kg/m2
* Willingness to give up being a blood donor from 4 weeks before the start of the study, during the study and for 4 weeks after completion of the study

Exclusion Criteria:

* Excessive caffeine use
* Major psychiatric/mental health disorders .
* Chronic sleep disorders
* Severe sleep disturbance for more than 1 year
* Other clear causes for poor sleep quality or mental wellbeing
* Use of medication or supplements that can affect outcomes
* Nonpharmacological treatment for sleep disorders
* Flight from a time-zone with >3 h difference ≤1 week before an intervention period
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study
* Use of pre-, pro- or synbiotics within 1 month prior to the start of the study
* Reported weight loss or weight gain of >3 kg in the month prior to pre-study screening
* Smoking
* Abuse of products
* Known allergy to citruses
* Known pregnancy or lactation

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in sleep quality scores between the intervention and placebo group | 8 weeks of intervention
  Measured by a sleep quality questionnaire (PSQI)
Changes in sleep quality between the intervention and placebo group | 8 weeks of intervention
  Measured using actigraphy

SECONDARY OUTCOMES:
Changes in mental wellbeing between the intervention and placebo group | 8 weeks of intervention
  Measured by mental wellbeing questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Principal Investigator — Maastricht University; Tanja Adam, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands